CLINICAL TRIAL: NCT03388567
Title: Evaluation of the Effects of a Drug With Fiscalized Substances Dispensation, Health Education and Pharmacovigilance Continuing Education Program in Community Pharmacies: Study Protocol for a Multicenter, Cluster-randomized Controlled Trial
Brief Title: Evaluation of the Effectiveness of a Continuing Education Program in Community Pharmacies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Pedro Amariles, Investigador principal, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0017102017MC
Record Dates: First submitted 2017-11-28; First posted 2018-01-03 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-04

CONDITIONS: Controlled Drug Dependence
Keywords: Dispensation; Health Education; Pharmacovigilance; Pharmacists
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: study protocol for a multicenter, cluster-randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Staff pharmacy whith intervention (Experimental): Staff pharmacy who will receive continuous education through technology and communication tools, as well as accompaniment and advice from a pharmaceutical chemist
  Interventions: Other: Staff pharmacy whith intervention
- Staff pharmacy without intervention (No Intervention): Staff pharmacy who will receive only pharmacy information

INTERVENTIONS:
Other: Staff pharmacy whith intervention — Pharmacists who will receive continuous education through technology and communication tools, as well as accompaniment and advice from a pharmaceutical chemist
  Arms: Staff pharmacy whith intervention

SUMMARY:
Preventable failures in the drug chain are related to Drugs Problems Related Use and are associated with medication errors (prescription, dispensing, administration or use by the patient or caregiver), including failures In the Medication Supply System (availability and quality).

The controlled drugs are those that contain substances regulated by international conventions on drug control. They are important in various fields of medicine, such as pain management, obstetric emergencies, mental disorders such as the treatment of substance dependence, psychiatry and neurology. It has been defined as abuse of drugs the improper use of these for non-medical purposes, and associated with the use without medical prescription, which can produce addiction or psychic or physical dependence.

DETAILED DESCRIPTION:
Experimental study with random assignment of the staff pharmacist of Pharmacies. The staff pharmacists admitted will be followed for 12 months (1 year). The study will make it possible to determine the effect of the continuing education program accompanied by Information and Communication Technologies (ICT).

ELIGIBILITY:
Inclusion Criteria:

1. Pharmacy staff working in Pharmacy or Drugstore, located geographically in the city of Medellín and in the Metropolitan Area
2. That the owner works in the establishment

Inclusion Exclusion:

1. Pharmacy staff who do not agree to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Pharmacy staff competences (Pharmacy staff knowledge, skills and attitudes. ) | 12 months
  Pharmacy staff knowledge, skills and attitudes.
  An adapted and self-designed questionnaire is used from different bibliographical references, among them, the General Level Framework (GLF), as well as the guidelines of the Colombian legislation for pharmacy staff competences. The main areas of competency (competency clusters): which are:
  * Delivery of patient care
  * Personal
  * Problem Solving
  * Management and Organisation
  The assessment rating is on a 4-point scale ranging from rarely, sometimes, usually to consistently:
  * Rarely: Very rarely meets the standard expected. No logical thought process appears to apply (0-20 %)
  * Sometimes: Much more haphazard than "usually" (21-50 %)
  * Usually: Implies standard practice with occasional lapses (51-84 %)
  * Consistently: Demonstrates the expected standard of practice with very rare lapses (85-100 %)

SECONDARY OUTCOMES:
Characterize the processes associated with the use of medications in the Pharmaceutical Establishments | 2 months
  Recognize basic information of the Pharmaceutical Establishments (PE), to characterize some processes related to the use of controlled drugs (CD), including compliance with the regulations, and determine the level of risk perception and the continuing education needs of the pharmacy staff. An adapted and self-designed questionnaire is used from different bibliographical references.
  The assessment rating is on a 4-point scale ranging from rarely, sometimes, usually to consistently:
  * Rarely: Very rarely meets the standard expected. No logical thought process appears to apply (0-20 %)
  * Sometimes: Much more haphazard than "usually" (21-50 %)
  * Usually: Implies standard practice with occasional lapses (51-84 %)
  * Consistently: Demonstrates the expected standard of practice with very rare lapses (85-100 %)
Implementation of pharmaceutical professional services | 12 months
  Measure the degree of implementation of pharmaceutical professional services: Dispensation, Health Education and Pharmacovigilance services. An adapted and self-designed questionnaire is used from different bibliographical references, among them, the guidelines of the Colombian legislation for the development of pharmaceutical services.
  The assessment rating is on a 4-point scale ranging from rarely, sometimes, usually to consistently:
  * Rarely: Very rarely meets the standard expected. No logical thought process appears to apply (0-20 %)
  * Sometimes: Much more haphazard than "usually" (21-50 %)
  * Usually: Implies standard practice with occasional lapses (51-84 %)
  * Consistently: Demonstrates the expected standard of practice with very rare lapses (85-100 %)
Satisfaction level pharmacy staff | 12 months
  Pharmacy staff satisfaction about the continuing education program. An adapted and self-designed questionnaire is used from different bibliographical references, among them, the General Level Framework (GLF), as well as the guidelines of the Colombian legislation for the development of labor competences from the pharmaceutical services.
  A five points scale (5=Excellent, 4=Good, 3=Satisfactory, 2=Needs Improvement, and 1=Unacceptable) will used in the questionnaire.
Satisfaction level patients | 12 months
  Patients satisfaction of pharmacy professional services. An adapted and self-designed questionnaire is used from different bibliographical references.
  A five points scale (5=Excellent, 4=Good, 3=Satisfactory, 2=Needs Improvement, and 1=Unacceptable) will used in the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Amariles, PhD, Principal Investigator — Universidad de Antioquia
Locations (1):
- Universidad de Antioquia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ceballos M, Salazar-Ospina A, Sabater-Hernandez D, Amariles P. Evaluation of the effects of a drug with fiscalized substance dispensation, health education, and pharmacovigilance continuing education program in Colombia drugstores and drugstores/pharmacies: study protocol of a multicenter, cluster-randomized controlled trial. Trials. 2020 Jun 19;21(1):545. doi: 10.1186/s13063-020-04481-1. PMID 32560735